CLINICAL TRIAL: NCT00370864
Title: Phase II Study of a Pandemic Influenza Vaccine in Children
Brief Title: Study of a Pandemic Influenza Vaccine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSLCT-PAN-05-17
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
Keywords: Pandemic; Influenza; Prevention; Vaccine; Prevention of Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: H5N1 pandemic influenza vaccine

SUMMARY:
The World Health Organisation has warned that an influenza pandemic is inevitable. The avian influenza strain H5N1 is one of the leading candidates to cause the next influenza pandemic. Children are likely to be a special target group for vaccination; therefore, this study will test the safety and immunogenicity of an H5N1 pandemic influenza vaccine in healthy children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged greater or equal to 6 months to less than 9 years
* Normal gestation period

Exclusion Criteria:

* History of clinically significant medical conditions
* History of Guillain Barre syndrome or active neurological disease

Ages: 6 Months to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2006-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Terry M Nolan, Prof, Principal Investigator — Murdoch Childrens Research Institute
Locations (2):
- Australia (2):
  - Murdoch Childrens Research Institute, Melbourne, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia

REFERENCES:
- [Derived] Nolan T, Richmond PC, Formica NT, Hoschler K, Skeljo MV, Stoney T, McVernon J, Hartel G, Sawlwin DC, Bennet J, Ryan D, Basser RL, Zambon MC. Safety and immunogenicity of a prototype adjuvanted inactivated split-virus influenza A (H5N1) vaccine in infants and children. Vaccine. 2008 Nov 25;26(50):6383-91. doi: 10.1016/j.vaccine.2008.08.046. Epub 2008 Sep 16. PMID 18801398